CLINICAL TRIAL: NCT01164280
Title: The Effect of Pulse Rate Changes on Clinical Outcome in Sacral Neuromodulation
Brief Title: Effect of Pulse Rate Changes on Clinical Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Philip van Kerrebroeck, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: MEC 07-2-083 (5266)
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Overactive Bladder Syndrome; Chronic Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulse Rate Change (Experimental): Patients are subjected to different pulse rate settings of their neurostimulator. The effect of pulse rate changes on clinical outcome is measured.
  Interventions: Other: Pulse Rate Change

INTERVENTIONS:
Other: Pulse Rate Change — Different pulse rate settings of the implantable neurostimulator

SUMMARY:
Objectives: To evaluate the effect of pulse rate changes on the clinical response and stimulation related pain symptoms in sacral neuromodulation (SNM) treatment.

Materials and Methods: This pilot study evaluated the effect of 4 different pulse rates (5.2Hz-10Hz-21Hz-40Hz) in patients with suboptimal response to SNM. The effect of each frequency was evaluated over test period of 6 days. To avoid carry over effect, stimulation was kept off for 24 hours between consecutive test periods. The last 3 days of every test period, a voiding diary (VD) and questionnaire was filled in. The changes on clinical response and pain symptoms were compared between the four pulse-rates using multivariate analysis.

Results: Fifty patients were included of which 40 (80%) were female. Mean age was 55.5yr (SD 12.3). Forty-one patients (82%) had overactive bladder symptoms and 9 (18%) had chronic non-obstructive urinary retention. No significant difference was found regarding clinical outcome (VD and questionnaire) between the different pulse rates. Furthermore, none of the four pulse rates was significantly related to the occurrence of SNM-related pain. However, on individual basis, patients appear to benefit from changing the pulse rate concerning both treatment efficacy and stimulation related pain.

Conclusions: On group level, none of the four pulse rates in this study appears to have a significantly different effect on clinical outcome or SNM-related pain. However, a tailor-made approach for optimizing treatment efficacy by changing the pulse rate might be useful.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been implanted with a neurostimulator for overactive bladder symptoms or urinary retention
* Patients with suboptimal effect of their neurostimulator

Exclusion Criteria:

* Patients with 100% effect of their neurostimulator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Improvement in voiding diary variables

SECONDARY OUTCOMES:
Improvement in subjective voiding symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Philip van Kerrebroeck, M.D., Ph.D., Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands